CLINICAL TRIAL: NCT02921217
Title: Randomized, Parallel, Double Blinded, Placebo-controlled Study for the Evaluation of the Effectiveness on Visceral Fat Accumulation in Individuals With Abdominal Obesity of a Specific Probiotic Compound
Brief Title: Effect of a Probiotic on Visceral Fat Accumulation
Acronym: BIFFAT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biopolis S.L. (Industry)
Collaborators: Technological Centre of Nutrition and Health (Other); Hospital Universitari Sant Joan de Reus (Other); University Rovira i Virgili (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BIFFAT
Record Dates: First submitted 2016-07-20; First posted 2016-10-03 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-09

CONDITIONS: Obesity; Intra-Abdominal Fat; Subcutaneous Fat, Abdominal
Keywords: Cardiovascular diseases; abdominal visceral fat; subcutaneous body fat; body weight; waist circumference; lipid profile; insulin resistance; glucose metabolism; blood pressure; inflammation; adiponectin; leptin; metabolomics; cardiovascular risk factor
MeSH Terms: conditions — Obesity; Cardiovascular Diseases; Body Weight; Insulin Resistance; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ActivBPL1 (Experimental): Active Probiotic Bifidobacterium animalis subsp. lactis BPL1 (CECT 8145)
  Interventions: Dietary Supplement: Active Probiotic
- InactivBPL1 (Experimental): Inactivated probiotic Bifidobacterium animalis subsp. lactis BPL1 (CECT 8145)
  Interventions: Dietary Supplement: Inactivated probiotic
- Control (Placebo Comparator): Control
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Active Probiotic — Product 1: 200 mg maltodextrin and 100 mg of active Bifidobacterium animalis subsp. lactis BPL1 (CECT 8145) (1011 CFU/g),
  Arms: ActivBPL1
Dietary Supplement: Inactivated probiotic — Product 1: 200 mg maltodextrin and 100 mg of Bifidobacterium animalis subsp. lactis BPL1 (CECT 8145) inactivated by heat (1011 CFU/g),
  Arms: InactivBPL1
Dietary Supplement: Control — Placebo: 300 mg maltodextrin.
  Arms: Control

SUMMARY:
The study's main objective is to investigate if an extract containing the probiotic Bifidobacterium animalis subsp. lactis BPL1 (CECT 8145) has a positive effect on the accumulation of abdominal visceral fat in people with abdominal obesity.

DETAILED DESCRIPTION:
The study's main objective is to investigate if an extract containing the probiotic Bifidobacterium animalis subsp. lactis BPL1 (CECT 8145) has a positive effect on the accumulation of abdominal visceral fat in people with abdominal obesity.

Participants: 129 men and women with a waist circumference ≥102 cm (men) or ≥88 cm (women), randomly assigned to one of 3 treatment groups in parallel: one group (43 members) with active probiotic, another one with the probiotic inactivated by heat, and the last group with the placebo.

Treatment consists of product consumption study for 12 weeks, taking 1 capsule per day. 4 visits during the study, a pre-inclusion visit and 3 study visits (weeks 1, 6, and 12) will be scheduled.

Secondary objectives are to asses the probiotic's effects on:

* the accumulation of subcutaneous body fat and body weight, body mass index (BMI) and waist circumference.
* glucose metabolism and insulin resistance.
* blood lipid profile.
* blood pressure.
* inflammation.
* circulating levels of adiponectin and leptin.
* changes in the intestinal microbiome

The statistical analysis will follow the principles specified in the guidelines of the ICHE9 and CPMP/EWP/908/99 ICHE9 Points to Consider on Multiplicity Issues in Clinical Trials.

ELIGIBILITY:
Inclusion Criteria:

* Adults men or women (>18 years old)
* Waist circumference ≥102 cm (men) or ≥88 cm (women) and <150cm
* Written informed consent provided before the initial screening visit.

Exclusion Criteria:

* Use of antibiotics within 30-days period before the study
* Waist circumference other than those specified in inclusion criteria
* Body mass index (BMI) ≥ 40 kg/m2
* Glucose (fasting state) ≥ 126 mg/dL
* Anemia (hemoglobin ≤13 g/dL in men and ≤12 g/dL in women)
* Suffer from claustrophobia (to the extent that precludes NMR).
* Wear pacemakers, electrical stimulators or cochlear implants (NMR contraindications)
* Following a hypocaloric diet and/or receiving pharmacologic treatment for weight loss
* Having eating disorders.
* Use of medication, antioxidant, or multi-vitamin supplements interfering with the study
* Chronic gastrointestinal pathology
* Being intolerant or suffer from allergy to any of the products of the study.
* Pregnant or intending to become pregnant
* Being in breastfeeding period.
* Chronic alcoholism
* Current or past participation in a clinical trial or consumption of a research product in the 30 days prior to inclusion in the study.
* Failing to follow study guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-05 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Change of abdominal visceral fat | Change from 0 weeks (V1) to 12 weeks (V3)
  abdominal visceral fat will be measured by Nuclear Magnetic Resonance (NMR). The study will be conducted in 3 Teslas MRI (Signa LX Echo Speed Plus Excite, General Electric, Milwaukee, WI).

SECONDARY OUTCOMES:
Change of body weight | Change from 0 weeks (V1) to 6 weeks (V2), and to 12 weeks (V3)
  Body weight measured with Tanita TBF-300 (Body Composition Analyzer, Brooklyn NY, USA)
Change of BMI | Change from 0 weeks (V1) to 6 weeks (V2), and to 12 weeks (V3)
  Calculated using weight and height. Body weight measured with Tanita TBF-300 (Body Composition Analyzer, Brooklyn NY, USA). Height, measured by Tanita portable altimeter; BMI calculated (kg/m2)
Change of Waist circumference | Change from 0 weeks (V1) to 6 weeks (V2), and to 12 weeks (V3)
  Waist circumference, measured according to the criteria of Lohman et al. 1988.
Change of Abdominal subcutaneous fat | Change from 0 weeks (V1) to 12 weeks (V3)
  Abdominal subcutaneous fat measured by 3 Teslas MRI (Signa LX Echo Speed Plus Excite, General Electric, Milwaukee, WI).

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Solà, Prof. MD, Principal Investigator — University Rovira i Virgili / Hospital Universitari Sant Joan de Reus
Locations (1):
- Technological Centre of Nutrition and Health (CTNS), Reus, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vaccaro O, Masulli M, Cuomo V, Rivellese AA, Uusitupa M, Vessby B, Hermansen K, Tapsell L, Riccardi G. Comparative evaluation of simple indices of insulin resistance. Metabolism. 2004 Dec;53(12):1522-6. doi: 10.1016/j.metabol.2004.05.017. PMID 15562393
- See also: Technological Centre of Nutrition and Health — http://www.ctns.cat